CLINICAL TRIAL: NCT05106361
Title: MOSAIC (MOthers' AdvocateS In the Community) for Pregnant Women and Mothers of Children Under 5 With Experience of Intimate Partner Violence: Randomized Trial
Brief Title: MOSAIC (MOthers' AdvocateS In the Community) for Pregnant Women and Mothers of Children Under 5 With Experience of Intimate Partner Violence
Acronym: MOSAIC Plus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Maji Debena, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 351185
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Intimate Partner Violence; Depression; Post Traumatic Stress Disorder
Keywords: Intimate partner violence; Women; Mothers; Pregnant
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic | interventions — Mosaicism

STUDY DESIGN:
Intervention Model Description: The proposed study will enroll pregnant women who report experience of IPV in the past 6 months, and who screen positive for elevated depressive and/or PTSD symptoms. The intervention lasts 9 months after enrollment. Those in the intervention arm will receive MOSAIC Plus (an enhanced MOSAIC intervention that includes IPT) while those in the active control would receive MOSAIC intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOSAIC Plus (Experimental): "Mother AdvocateS In the Community (MOSAIC) Plus" intervention to reduce depressive and PTSD symptoms and prevent additional IPV among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate IPT principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms.
  Interventions: Behavioral: MOSAIC Plus
- MOSAIC (Active Comparator): Those in the active comparator will receive the "Mother AdvocateS In the Community (MOSAIC) Plus" intervention to reduce depressive and PTSD symptoms and prevent additional IPV among pregnant women and mothers with children under 5 experiencing IPV.
  Interventions: Behavioral: MOSAIC

INTERVENTIONS:
Behavioral: MOSAIC Plus — Those in the experimental arm will receive the intervention is called "Mother AdvocateS In the Community (MOSAIC) Plus", an intervention to reduce depressive and PTSD symptoms and prevent additional intimate partner violence among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate interpersonal psychotherapy principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms.
  Arms: MOSAIC Plus
Behavioral: MOSAIC — Those in the active comparator will receive a mentor mother intervention named Mother AdvocateS In the Community (MOSAIC). This does not include the IPT component.
  Arms: MOSAIC

SUMMARY:
The purpose of this R34 exploratory research proposal is to conduct formative work for a larger randomized controlled trial (RCT) evaluating the effectiveness of the "Mother AdvocateS In the Community (MOSAIC) Plus" intervention to reduce depressive and PTSD symptoms and prevent additional IPV among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate IPT principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms. The proposed study will enroll pregnant women who report experience of IPV in the past 6 months, and who screen positive for elevated depressive and/or PTSD symptoms. The intervention lasts 6 months after enrollment.

DETAILED DESCRIPTION:
Violence against women is a global human rights concern and a significant public health challenge; 1 in 3 three women experience lifetime physical and/or sexual violence.1 As many as 5.3 million U.S. women report experiencing intimate partner violence (IPV; referring to sexual or physical violence by current or former partners) annually2. Depression and posttraumatic stress disorder (PTSD) are the two most common mental health consequences of IPV. In turn, developing depressive and PTSD symptoms after experiencing IPV increases future risk of IPV3. IPV is also associated with chronic physical health problems4,5 and self-harm 6.

Motherhood and pregnancy increase the risk for prolonged exposure to physical, psychological and sexual IPV7. With as many as 4% to 8% of pregnant women reporting IPV during pregnancy, IPV can start or worsen during the perinatal period8. Previous and current experience of IPV is strongly associated with poor physical health, mental health and obstetric outcomes9,10; leading to increased utilization of health services11 even after the IPV ends12. There are very few interventions that effectively reduce IPV among pregnant women and mothers with children under 5 who report IPV13-15. One of them, Mother AdvocateS In the Community (MOSAIC) forms the basis of this proposal16. No existing intervention addresses the depressive and PTSD symptoms that often follow IPV, are associated with suffering and morbidity, and potentiate future IPV risk for pregnant women and mothers with children under 5 who report IPV. In fact, there are not any interventions for any group of women that effectively reduce both future IPV risk and common related mental health symptoms such as depression and PTSD. An integrated intervention that addresses elevated symptoms of maternal depression and PTSD while reducing subsequent IPV is needed.

MOSAIC is a non-professional intervention delivered by mentor mothers from the community to reduce IPV in pregnant women and mothers with children under 517. The intervention combines elements of mentoring and IPV-specific support provided by mentor mothers. MOSAIC was also tested in a fully-powered RCT for pregnant women and mothers with children under 5 in Australia and found to reduce subsequent IPV15. However, it did not significantly improve depression, and PTSD symptoms were not evaluated. Given the suffering, morbidity, and additional risk of IPV conferred by depressive and PTSD symptoms, the proposed study will augment MOSAIC with principles of an evidence-based intervention to improve maternal mental health. Interpersonal psychotherapy (IPT) is the front-line treatment for maternal depression18 and has been found to reduce PTSD symptoms in the perinatal period19. IPT addresses maternal mental health by helping women increase their general social support systems and build communication skills and confidence to access needed resources and help. IPT can be effectively delivered by lay providers. This proposal will integrate IPT principles into MOSAIC to address both IPV and its mental health sequelae.

The purpose of this R34 exploratory research proposal is to conduct formative work for a larger randomized controlled trial (RCT) evaluating the effectiveness of the "Mother AdvocateS In the Community (MOSAIC) Plus" intervention to reduce depressive and PTSD symptoms and prevent additional IPV among pregnant women and mothers with children under 5 experiencing IPV. The MOSAIC Plus intervention will integrate IPT principles and skills into the MOSAIC intervention in order to expand it to address consequences of IPV, including depression and PTSD symptoms. The proposed study will enroll pregnant women who report experience of IPV in the past 6 months, and who screen positive for elevated depressive and/or PTSD symptoms. The intervention lasts 9 months after enrollment. Women will be recruited from Obstetrics and Gynecological unit of the Hurley Medical Center and YWCA, Flint. The control condition will be the original MOSAIC intervention. Study assessments will take place at baseline, 3, 6 and 9 months.

The development aims of this proposal are to:

1. Enhance and expand the MOSAIC manual (designed to be delivered by lay providers) with lay-provider friendly IPT principles for reducing depressive and PTSD symptoms.
2. Refine the manual, intervention, and study procedures using 6 focus groups: 3 groups with mothers who have experienced IPV in the past 6 months (n~20), 2 with potential mentor mothers (n~16), and 1 group with nurse-family partnership staff (n~8)
3. Develop, implement, and evaluate the intervention training program.
4. Improve the clarity, content, acceptability, and feasibility of the enhanced MOSAIC Plus intervention through a small open trial (n = 15) of mothers with past 6-month IPV experience

   The pilot study aims of this proposal are to:
5. Conduct a pilot RCT in a sample of 40 mothers with IPV experience in the past 6 months to demonstrate the feasibility and acceptability of the proposed recruitment methods, research design, intervention training methods, and of delivering the MOSAIC Plus and MOSAIC interventions. As recommended by NIMH, we will also examine 95% confidence intervals around differences between the proposed intervention and MOSAIC for the following outcomes through 9 months after baseline:

   1. Mental health outcomes. Reduction in depressive (primary) and PTSD symptoms
   2. IPV outcomes. Decreased subsequent IPV over the 9 months measured by CAS
   3. Functioning outcomes. Improvement in functioning, self-care and general health and wellbeing
   4. Potential target mechanisms. Increased social support and effectiveness obtaining resources.

Interventions to improve mental health challenges experienced by mothers who experienced IPV are of great public health significance. Reducing depressive and PTSD symptoms in women with the experience of IPV has significant public health benefits for mothers and their children.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and/or are mothers of children under 5 and r
* Report IPV experiences in the past 6 months (as assessed by Composite Abuse Scale)
* Aged 18 or above,
* Have elevated depressive and/or PTSD symptoms as assessed by Patient Health Questionnaire (PHQ-9) with a cutoff point of ≥9, and/or the Davidson Trauma Scale (DTS) with a cut-off point of ≥40.

Exclusion Criteria:

* Cannot provide the name and contact information of at least two locator persons,
* Do not have access to any telephone,
* Cannot understand English well enough to understand the consent form or assessment instruments when they are read aloud

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
acceptability | 9 months
  We will evaluate the acceptability of the proposed recruitment methods, research design, intervention training methods, and of delivering the MOSAIC Plus and MOSAIC interventions by using End of Treatment Questionnaire.
Satisfaction with care | 9 months
  We will evaluate the feasibility of the proposed recruitment methods, research design, intervention training methods, and of delivering the MOSAIC Plus and MOSAIC interventions by using Client Satisfaction Questionnaire.
Quality of Working Relationship | 9 months
  We will evaluate therapeutic alliance by using Working Alliance Inventory-Short Revised (WAI-SR)
Reduction in depressive symptoms | baseline, 3, 6 and 9 months
  We will measure reduction in depressive symptoms as assessed by Patient Health Questionnaire (PHQ-9).
Reduction in Posttraumatic Stress Disorder Symptoms | baseline, 3, 6 and 9 months
  We will measure reduction in posttraumatic stress disorder symptoms by using Davidson Trauma Scale.

SECONDARY OUTCOMES:
Intimate Partner Violence | baseline, 3, 6 and 9 months
  We will measure reduction in subsequent intimate partner violence by using Composite Abuse Scale.
Effectiveness Obtaining Resources | baseline, 3, 6 and 9 months
  We will measure effectiveness in obtaining resources by using Effectiveness Obtaining Resources (EOR) scale.
Perceived Social Support | baseline, 3, 6 and 9 months
  We will measure improvements in perceived social support by using The RAND social support scale (Medical Outcome Study-Social Support Survey MOS-SS)
Functioning | baseline, 3, 6 and 9 months
  We will use the WHO Disability Assessment schedule-12 to assess mental health related disability.
Self-care and self-worth | baseline, 3, 6 and 9 months
  We will use the self-care and self-worth scale to assess changes in self-care.
General health and wellbeing | baseline, 3, 6 and 9 months
  We will use the SF-36 to assess changes in general health and wellbeing.

OTHER OUTCOMES:
Provider Competencies | 6 and 9 months
  We will assess competency of providers by using Competency Assessment Inventory (CAI)
Quality of working relationship-provider perspective | 3, 6 and 9 months
  We will assess the quality of working relationship by using the provider perspective section of working alliance inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- YWCA Flint, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided